CLINICAL TRIAL: NCT05261347
Title: Effect of Mulligan Movement Mobilization Technique on Elbow Joint Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Kevser Sevik, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DokuzEU131313
Record Dates: First submitted 2021-12-05; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Healthy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): mobilisation group
  Interventions: Procedure: mulligan mobilisation
- control (Sham Comparator): sham control group
  Interventions: Procedure: sham

INTERVENTIONS:
Procedure: mulligan mobilisation — an active mobilisation with movement on elbow according to mulligan's protocol
  Arms: intervention
Procedure: sham — a lateral glide
  Arms: control

SUMMARY:
Investigating The Effects of Mulligan Movement Mobilization Technique on Elbow Joint Proprioception

DETAILED DESCRIPTION:
Investigating The Effects of Mulligan Movement Mobilization Technique on Elbow Joint Proprioception by joint position sense assessment

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years

Exclusion Criteria:

* having any elbow condition
* having any neurological condition

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
elbow proprioception assessment by evaluating joint position sense | 35 minutes
  joint position sense error measurement with universal goniometer at 70 and 110 degrees of flexion

CONTACTS AND LOCATIONS:
Overall Officials: kevser sevik, Principal Investigator — Dokuz Eylul University
Locations (1):
- Physical Therapy and Rehabilitation School, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevik Kacmaz K, Unver B. Immediate Effects of Mulligan Mobilization on Elbow Proprioception in Healthy Individuals: A Randomized Placebo-Controlled Single-Blind Study. J Manipulative Physiol Ther. 2023 Jan;46(1):59-64. doi: 10.1016/j.jmpt.2023.05.001. Epub 2023 Jul 7. PMID 37422752